CLINICAL TRIAL: NCT03896659
Title: Exploring the Effects of Corticosteroids on the Human Hippocampus Using Neurocognitive Testing and High Resolution Neuroimaging
Brief Title: Exploring the Effects of Corticosteroids on the Human Hippocampus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, Irvine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU-2018-0360; 1R01MH115932-01A1 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hydrocortisone; Depression; Healthy Volunteers
MeSH Terms: conditions — Depression | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Depressed: Hydrocortisone, then Placebo (Experimental): Participants in the "depressed' arm will receive a Hydrocortisone 160 mg tablet every day for 3 days. After a washout period of 25 days, they then will receive a Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days.
  Interventions: Drug: Hydrocortisone Oral; Drug: Placebo Oral Tablet
- Depressed: Placebo, then Hydrocortisone (Experimental): Participants in the "depressed' arm will receive a Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days. After a washout period of 25 days, they then will receive a Hydrocortisone 160 mg tablet every day for 3 days.
  Interventions: Drug: Hydrocortisone Oral; Drug: Placebo Oral Tablet
- Healthy Controls: Hydrocortisone, then Placebo (Experimental): Participants in the "healthy control" arm will receive a Hydrocortisone 160 mg tablet every day for 3 days. After a washout period of 25 days, they then will receive a Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days.
  Interventions: Drug: Hydrocortisone Oral; Drug: Placebo Oral Tablet
- Healthy Controls: Placebo, then Hydrocortisone (Experimental): Participants in the "healthy control" arm will receive a Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days. After a washout period of 25 days, they then will receive a Hydrocortisone 160 mg tablet every day for 3 days.
  Interventions: Drug: Hydrocortisone Oral; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Hydrocortisone Oral — Hydrocortisone 160 mg tablet
Drug: Placebo Oral Tablet — Hydrocortisone-matched Placebo tablet

SUMMARY:
Chronic corticosteroid (CS) exposure is associated with changes in memory and the hippocampus in both humans and in animal models. The hippocampus has a high concentration of glucocorticoid receptors (GCRs), and the pre-clinical literature demonstrates shortening of apical dendrites in the CA3 region of the hippocampus and decreased neurogenesis in the dentate gyrus (DG) following CS administration. In humans, both stress and CS exposure are associated with a decline in declarative memory performance (a process mediated by the hippocampus). Impairment in declarative memory and hippocampal atrophy are reported in patients with excessive CS release due to Cushing's disease, and, by our group, in patients receiving prescription CS therapy. These findings have important implications for patients with mood disorders, as a large subset of people with major depressive disorder (MDD) show evidence of HPA axis activation, elevated cortisol and, importantly, resistance to the effects of CSs on both the HPA axis and on declarative memory. Thus, resistance to corticosteroids appears to be a consequence of MDD.

this study will examine changes in declarative memory, as well as use state-of-the-art high-resolution multimodal neuroimaging, including structural and functional (i.e., task-based and resting state) MRI, in both men and women healthy controls, and, as an exploratory aim, a depressed group, given 3-day exposures to hydrocortisone (160 mg/day) or placebo. The study will translate preclinical findings to humans, provide valuable data on possible sex differences in the response to cortisol and, for the first time, identify specific hippocampal subfields (e.g., CA3/DG) in humans that are most sensitive to acute CS effects. Using resting state fMRI data and whole brain connectomics using graph theoretical approaches, we will determine the effects of cortisol exposure on functional brain networks. Furthermore, this will be the first study to use neuroimaging to compare the brain's response to CSs in people with depression vs. controls, and determine whether depressed people demonstrate glucocorticoid resistance within the hippocampus. We hypothesize that hippocampal response to acute CSs will be greatest in the CA3/DG subfield, greater in women than in men, and that depressed people will show a blunted hippocampal response to CSs compared to controls. A multidisciplinary research team with extensive experience in CS effects on the brain and hippocampal subfield neuroimaging, and a prior history of research collaboration, will conduct the project.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-50 years with vision corrected to at least 20-40 (needed for fMRI tasks)
* Education of ≥ 12 years
* Baseline RAVLT total words recalled T-score ≥ 40 (normal range)
* BMI between 18.5-35.0 (neither underweight nor severely obese)
* Baseline QIDS-C ≤ 5 (virtual absence of depressive symptoms) for "healthy controls" and for the "depressed" group a QIDS-C between 11-20 (≥ moderate depressive symptoms but < very severe depressive symptoms)

Exclusion Criteria:

* History of major psychiatric illness other than MDD for the depressed group, defined as bipolar disorder, posttraumatic stress disorder, schizoaffective disorder, schizophrenia, eating disorders, or MDD with psychotic features. For the control group, a past episode of MDD (per SCID) is also exclusionary
* History of drug or alcohol use disorder
* History of neurological disorders including seizures, brain surgery, multiple sclerosis, Parkinson's disease
* Taking CNS-acting medications (e.g., antidepressants, antipsychotics, lithium, anticonvulsants, sedative/hypnotic/anxiolytics). Thus, the depressed group will be medication free.
* History of allergic reaction or medical contraindication to hydrocortisone
* Metal implants, claustrophobia, or other contraindications to MRI
* Significant medical conditions (e.g., cancer, heart disease, diabetes)
* Vulnerable population including pregnant or nursing women, prisoners, and people with intellectual disability, history of special education classes, dementia, or other severe cognitive disorders
* Current suicidal ideation, a suicide attempt in the past 12 months or more than one lifetime attempt
* History of systemic CS use in the past 12 months, lifetime cumulative use of more than 12 weeks, or recent (defined as past 28 days) inhaled CS use
* Women who are using estrogen containing oral contraceptive agents (other contraceptives are acceptable, see Protection of Human Subjects section for a list of acceptable birth control methods) or who are post- or peri-menopausal or with irregular menstrual cycles (i.e., inconsistent menstruation patterns)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants included healthy controls and adults with depression being treated at UT Southwestern Medical Center.
Groups:
- Depressed: Hydrocortisone, Then Placebo: Participants in the "Depressed' arm first received Hydrocortisone 160 mg tablet every day for 3 days. After a washout period of 25 days, they then received a Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days.
- Depressed: Placebo, Then Hydrocortisone: Participants in the "Depressed' arm first received Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days. After a washout period of 25 days, they then received Hydrocortisone 160 mg tablet every day for 3 days.
- Healthy Controls: Hydrocortisone, Then Placebo: Participants in the "Healthy Controls' arm first received Hydrocortisone 160 mg tablet every day for 3 days. After a washout period of 25 days, they then received a Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days.
- Healthy Controls: Placebo, Then Hydrocortisone: Participants in the "Healthy Controls' arm first received Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days. After a washout period of 25 days, they then received Hydrocortisone 160 mg tablet every day for 3 days.
Period: First Intervention (3 Days)
Arm/Group | Depressed: Hydrocortisone, Then Placebo | Depressed: Placebo, Then Hydrocortisone | Healthy Controls: Hydrocortisone, Then Placebo | Healthy Controls: Placebo, Then Hydrocortisone
Started | 12 | 11 | 22 | 21
Completed | 12 | 9 | 20 | 21
Not Completed | 0 | 2 | 2 | 0
Period: Washout (25 Days)
Arm/Group | Depressed: Hydrocortisone, Then Placebo | Depressed: Placebo, Then Hydrocortisone | Healthy Controls: Hydrocortisone, Then Placebo | Healthy Controls: Placebo, Then Hydrocortisone
Started | 12 | 9 | 20 | 21
Completed | 10 | 7 | 16 | 20
Not Completed | 2 | 2 | 4 | 1
Period: Second Intervention (3 Days)
Arm/Group | Depressed: Hydrocortisone, Then Placebo | Depressed: Placebo, Then Hydrocortisone | Healthy Controls: Hydrocortisone, Then Placebo | Healthy Controls: Placebo, Then Hydrocortisone
Started | 10 | 7 | 16 | 20
Completed | 8 | 7 | 16 | 19
Not Completed | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depressed: Hydrocortisone, Then Placebo | Depressed: Placebo, Then Hydrocortisone | Healthy Controls: Hydrocortisone, Then Placebo | Healthy Controls: Placebo, Then Hydrocortisone | Total
Number analyzed (Participants) | 12 | 11 | 22 | 21 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 22 | 21 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.25 (11.07) | 41.73 (8.57) | 29.45 (9.26) | 31.00 (9.36) | 32.50 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 14 | 10 | 42
  Male | 3 | 2 | 8 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 4 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 2 | 2 | 10
  White | 8 | 5 | 14 | 15 | 42
  More than one race | 2 | 0 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 8 | 9 | 22
  Not Hispanic or Latino | 9 | 9 | 14 | 10 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Hippocampal Subfield Activation (Left Hemisphere)
Description: The z-scores of hippocampal subregions and hemispheres represent the standardized difference in activation between correct and incorrect conditions of the mnemonic discrimination task, where a Z-score of 0 represents the mean difference across all voxels, and each unit reflects one standard deviation from that mean. To compare brain activation between conditions, separate beta weights were estimated for correct and incorrect trials across all trials. These beta weights represent the voxel-wise blood oxygen level (BOLD)-dependent signal, reflecting changes in neural activity associated with each condition. Positive z-scores indicate greater activation for correct relative to incorrect trials, whereas negative z-scores indicate greater activation for incorrect relative to correct trials. Larger absolute z-scores indicate stronger condition-related effects; there are no established clinical thresholds for these experimental activation differences.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- Depressed: Hydrocortisone: Participants in the "Depressed' arm who received Hydrocortisone 160 mg tablet every day for 3 days as the first or second intervention.
- Depressed: Placebo: Participants in the "Depressed' arm who received Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days as the first or second intervention.
- Healthy Controls: Hydrocortisone: Participants in the "Healthy Controls' arm first received Hydrocortisone 160 mg tablet every day for 3 days as the first or second intervention.
- Healthy Controls: Placebo: Participants in the "Healthy Controls' arm first received Placebo tablet (matching Hydrocortisone 160 mg tablet) every day for 3 days as the first or second intervention.
Arm/Group | Depressed: Hydrocortisone | Depressed: Placebo | Healthy Controls: Hydrocortisone | Healthy Controls: Placebo
Number analyzed (Participants) | 13 | 11 | 15 | 16
Z-Score | -0.35 (0.76) | 0.03 (0.25) | -0.08 (0.57) | -0.07 (0.53)

2. Primary Outcome: Hippocampal Subfield Activation (Right Hemisphere)
Description: as for outcome 1
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Depressed: Hydrocortisone | Depressed: Placebo | Healthy Controls: Hydrocortisone | Healthy Controls: Placebo
Number analyzed (Participants) | 13 | 11 | 15 | 16
Z-Score | -0.05 (0.47) | -0.04 (0.41) | -0.09 (0.50) | -0.24 (0.37)

3. Primary Outcome: Hippocampal Subfield Volume (Left Hemisphere)
Description: High resolution structural neuroimaging will be used to generate regional hippocampal subfield volume.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Cubic Millimeter
Arm/Group | Depressed: Hydrocortisone | Depressed: Placebo | Healthy Controls: Hydrocortisone | Healthy Controls: Placebo
Number analyzed (Participants) | 18 | 17 | 36 | 33
Cubic Millimeter | 56.05 (15.67) | 54.65 (13.90) | 54.52 (12.43) | 50.55 (13.78)

4. Primary Outcome: Hippocampal Subfield Volume (Right Hemisphere)
Description: High resolution structural neuroimaging will be used to generate regional hippocampal subfield volume.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Cubic Millimeter
Arm/Group | Depressed: Hydrocortisone | Depressed: Placebo | Healthy Controls: Hydrocortisone | Healthy Controls: Placebo
Number analyzed (Participants) | 18 | 17 | 36 | 33
Cubic Millimeter | 65.95 (20.29) | 66.10 (20.68) | 65.65 (16.38) | 62.03 (17.08)

ADVERSE EVENTS:
Time Frame: The period of observation for the collection of adverse events extended from the time the subject gave informed consent until study completion, an average of 40 days.
Arm/Group | Depressed: Hydrocortisone | Depressed: Placebo | Healthy Controls: Hydrocortisone | Healthy Controls: Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/42 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/21 | 0/42 | 0/37
Other Adverse Events (participants affected / at risk) | 3/19 | 3/21 | 6/42 | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depressed: Hydrocortisone (N=19) | Depressed: Placebo (N=21) | Healthy Controls: Hydrocortisone (N=42) | Healthy Controls: Placebo (N=37)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depressed: Hydrocortisone (N=19) | Depressed: Placebo (N=21) | Healthy Controls: Hydrocortisone (N=42) | Healthy Controls: Placebo (N=37)
Daytime Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmares (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Difficulty Sleeping (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flushing in Face (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Burning Sensation in Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MRI Abnormality (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased Energy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loose Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne Exacerbation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema Flare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Racing Thoughts (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever Blister (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03896659/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03896659/ICF_001.pdf